CLINICAL TRIAL: NCT01152346
Title: A Multi-Center Relative Bioavailability Study of Azacitidine 75 mg/m2 Subcutaneous Injection In Myelodysplastic Syndrome Patients Under Fasting Conditions
Brief Title: Bioequivalence Study of Azacitidine for Injection in Myelodysplastic Syndrome (MDS) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bioniche Pharma USA LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AZFAST101
Record Dates: First submitted 2010-06-25; First posted 2010-06-29 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Myelodysplastic Syndrome
Keywords: Bioequivalence; Myelodysplastic Syndrome; MDS; Azacitidine
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ARM 1 (Other): Sequence- Azacitidine followed by Vidaza®
  Interventions: Drug: Azacitidine for Injection; Drug: Vidaza®
- ARM 2 (Other): Sequence-Vidaza® followed by Azacitidine
  Interventions: Drug: Azacitidine for Injection; Drug: Vidaza®

INTERVENTIONS:
Drug: Azacitidine for Injection — 75 mg/m2 sc injection on Day 1 of either cycle 1 or cycle 2 per randomization assignment
Drug: Vidaza® — 75 mg/m2 sc injection on Day 1 of either cycle 1 or cycle 2 per randomization assignment

SUMMARY:
The purpose of the study is to determine the bioavailability of Azacitidine for Injection relative to Vidaza® in MDS patients under fasting conditions. The data will be evaluated statistically to determine if the products meet bioequivalence criteria.

DETAILED DESCRIPTION:
This study is an open label, multi-center randomized, single dose, two-treatment, two-period, two-sequence, two-way cross-over, relative bioavailability study of Azacitidine for Injection for suspension use manufactured for Bioniche Pharma USA LLC compared with Vidaza® manufactured by Celgene Corporation in MDS patients under fasting conditions. Patients who are on a stable 75 mg/m2 dose of Vidaza will be randomized to study drug sequence Azacitidine on C1D1/ Vidaza® on C2D1 or Vidaza® on C1D1 / Azacitidine on C2D1. Randomization will be in a 2:2 ratio. Thirty-six (36) patients will be enrolled to ensure 28 evaluable patients. Patients will not be blinded to their treatment assignment.

After randomization, fasted patients will receive 1 dose of assigned study drug (either Azacitidine for Injection or Vidaza®) subcutaneously at a dose of 75 mg/m2 on C1D1. On Days 2-7, they will receive their normal Vidaza® treatment. Following a 21 day rest period, patients will cross over to receive the alternate treatment on C2D1 followed by their normal Vidaza®) treatment on Cycle 2 Days 2-7. The Final Patient Visit will be conducted 7 days following the last dose of Vidaza®.

The total duration of the study for each patient will be up to 56 days including the Screening period and Post Study Visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients with age >18 years.
* Patients with Myelodysplastic Syndrome (MDS) placed on Vidaza® according to the Marketing Authorization issued in the country in which the clinical study is being conducted (i.e., in the US, patients with any of the following French-American-British ( FAB) subtypes: Refractory Anemia (RA), Refractory Anemia with Ringed Sideroblasts (RARS), (if accompanied by neutropenia or thrombocytopenia or requiring transfusions), Refractory Anemia with Excess Blasts (RAEB), Refractory Anemia with Excess Blasts in Transformation (RAEB-T) and Chronic Myelomonocytic Leukemia (CMMoL); in France, subjects who are not eligible for hematopoietic stem cell transplantation: with intermediate -2 and high-risk myelodysplastic syndromes according to the International Prognostic Scoring System (IPSS) or chronic myelomonocytic leukemia (CMML) with 10-29% marrow blasts without myeloproliferative disorder) and who currently receive Vidaza at 75 mg/m2;
* Patient life expectancy > 6 months.
* Patients with performance status of 0 - 2 as per ECOG Scale.
* Patients with Total Bilirubin < 1.5 x ULN; ALT/AST < 2 x ULN, Serum Creatinine < 1.5 ULN, Serum Bicarbonate > 19 mEq/L.
* Patients who have signed the Informed Consent Form.

Exclusion Criteria:

* Patients with a history of alcoholism or drug addiction (during past 2 years)
* Patients with severe hepatic impairment, impaired renal function, and any condition which in the Investigator's opinion would be contraindicated or would interfere with absorption of the study drug.
* Patients whose clinical laboratory test values are outside the reference range may be re-tested at the discretion of the Investigator. If the clinical values are outside the range on re-testing, the patient will not be eligible to participate in the study unless the Investigator deems the result not to be significant.
* Patients with any other active malignancy within the past 5 years except for cervical cancer in situ, in situ carcinoma of the bladder or non-melanoma carcinoma of the skin.
* Patients who have a history of allergic responses to the class of drug being tested.
* Patients with hypersensitivity to Mannitol.
* Patients should not have donated blood and/or plasma for at least thirty (30) days prior to the first dosing of the study drug. Patients should not have had any transfusion of blood products for at least 7 days prior.
* Patients who have taken any investigational drug within thirty (30) days prior to the first dosing of the study.
* Female patients who are pregnant, breast-feeding, or who are likely to become pregnant during the study. Female patients of child bearing potential will be instructed to either abstain from sexual intercourse or use an acceptable method of birth control during the course of the study and for 3 months afterward. Male patients or their female partners should also use an acceptable method of birth control.
* Any patient whom the Investigator believes will not be a good candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Measurement of Azacitidine in Plasma Samples for Determination of Cmax, AUC0-t, and AUC0-Inf | 13 timepoints from pre-dose to 8 hours post dose
  Pharmacokinetic samples will be collected pre-dose and at 12 timepoints post-dose for determination of the level of azacitidine. The relative bioavailability of test to reference drug will be evaluated. If the Cmax, AUC0-t and AUC0-inf 90% confidence intervals for the geometric mean ratio all lie within 80-125% for Azacitidine then bioequivalence is concluded.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Throughout study
  Safety will be assessed through monitoring of adverse events and laboratory measures.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre FENAUX, MD Professor, Study Chair — Service d'hématologie clinique- Hôpital Avicenne; Emmanuel GYAN, MD, Principal Investigator — Centre régional de cancérologie Henry-Kaplan Service d'Hématologie et thérapie cellulaire-Hôpital Bretonneau; Agnès-Paule GUERCI-BRESLER, MD, Principal Investigator — Service d'hématologie et de médecine interne-Hôpital de Brabois; Jean-Richard Eveillard, MD, Principal Investigator — CHU de Brest- Hôpital Morvan; Odile BEYNE-RAUZY, MD Professor, Principal Investigator — University Hospital, Toulouse; Laurence LEGROS, MD, Principal Investigator — Hôpital Archet 1; Mauricette MICHALLET, MD Professor, Principal Investigator — Hôpital Edouard Herriot; Krimo Bouabdallah, MD, Principal Investigator — Hôpital Haut-Lévêque; Pascal Cony-Makhoul, MD, Principal Investigator — CH Annecy; Manjesh Lingamurthy, MD, Principal Investigator — Holy Cross Hospital; Steven Hager, MD, Principal Investigator — California Cancer Associates; Misagh Karimi, MD, Principal Investigator — Wilshire Oncology Medical Group; Veena Charu, MD, Principal Investigator — Pacific Cancer Medical Center Inc.
Locations (13):
- United States (4):
  - Pacific Cancer Medical Center Inc., Anaheim, California
  - Wilshire Oncology Medical Group, Corona, California
  - California Cancer Associates, Fresno, California
  - Holy Cross Hospital, Fort Lauderdale, Florida
- France (9):
  - Service d'hématologie clinique Hôpital Avicenne, Bobigny
  - CHU de Brest- Hôpital Morvan, Brest
  - Centre Hospitalier Lyon Sud, Lyon
  - Hôpital Archet 1, Nice
  - Hôpital Haut-Lévêque, Pessac
  - CH Annecy, Pringy
  - CHU Purpan, Toulouse
  - Centre régional de cancérologie Henry-Kaplan Service d'Hématologie et thérapie cellulaire, Tours
  - Service d'hématologie et de médecine interne CHU de Nancy Hôpital de Brabois, Vandœuvre-lès-Nancy